CLINICAL TRIAL: NCT04115722
Title: Coagulation Parameters in IBD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Mahmoud Hammam, Doctor, Assiut University
Other Study IDs: Coagulation parameters in IBD
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Agroup of IBD patients in activity
  Interventions: Other: IBD ACTIVIT
- Normal controlled group

INTERVENTIONS:
Other: IBD ACTIVIT — Effect of IBD disease and activity of disease on coagulation parameters
  Groups: Agroup of IBD patients in activity

SUMMARY:
1. to assess the incidence of coagulation disorders in IBD patients in comparison with another normal controlled group
2. risk factors that contribute to development of thrombosis in IBD patients
3. to determine the effectiveness of prophlactive anticoagulant measures
4. to determine the association between disease activity and coagulation parameters

DETAILED DESCRIPTION:
Inflammatory bowel disease is a group of disorders associated with chronic, recurrent, and immune system-mediated inflammation of The bowel mucosa . The reported global incidence and prevalence rates for ulcerative colitis vary between 1.2-20.3 and 6-246 per 100000 persons, respectively, and the corresponding figures for Crohns disease are 0.03-15.6 and 3.6-214 [2 In a population based cohort study involving 1160 patients with ulcerative colitis, the complication-related mortality rate was 9.6% during follow-up period of 35 years, in another study, 221 patients with Crohns disease were followed up for 33 years, with an overall complication-related mortality rate of Of the extra-intestinal manifestations of inflammatory bowel disease (IBD), thromboembolic events represent a major cause of morbidity and mortality with a 3.6 times increased risk in comparison with the general population .

Although clinical observations suggest an incidence rate between 1 and 8% for thromboembolic events in subjects with IBD, postmortem studies point out to a much higher occurrence rate around 41% . As a matter of fact, these and similar findings have led to an increased interest in the search for the association between IBD and hypercoagulable states as a potential cause of increased morbidity and mortality due to thromboembolic events in IBD . For instance, the existence of documentable prothrombotic abnormalities and a positive history for thromboembolic complications were demonstrated in at least one third of the subjects with IBD in a study by Solem et al Inflammation and coagulation are two crucial systems that are in balance and constantly influence each other. The impact of inflammation on coagulation has been confirmed by several experimental studies showing that inflammatory mechanism shift the hemostatic balance to favor the activation of coagulation which, in turn, can also sustain inflammation promoting a vicious circle between chronic inflammation and thrombosis

ELIGIBILITY:
Inclusion Criteria:

All patients of IBD more than 18 years

Exclusion Criteria:

-All IBD patients less than 18 years-all diseases that cause coagulation disorders all diseases that cause coagulation disorders ( liver diseases , collagen diseases, other auto immune disease

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study will be done on IBD patients espesially in activity to determine effect of disease on coagulation system
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of IBD patients in activity with DVT | Within one year dollow up

REFERENCES:
- [Background] Dolapcioglu C, Soylu A, Kendir T, Ince AT, Dolapcioglu H, Purisa S, Bolukbas C, Sokmen HM, Dalay R, Ovunc O. Coagulation parameters in inflammatory bowel disease. Int J Clin Exp Med. 2014 May 15;7(5):1442-8. eCollection 2014. PMID 24995109
- [Background] Sartor RB. Mechanisms of disease: pathogenesis of Crohn's disease and ulcerative colitis. Nat Clin Pract Gastroenterol Hepatol. 2006 Jul;3(7):390-407. doi: 10.1038/ncpgasthep0528. PMID 16819502
- [Background] Loftus EV Jr. Clinical epidemiology of inflammatory bowel disease: Incidence, prevalence, and environmental influences. Gastroenterology. 2004 May;126(6):1504-17. doi: 10.1053/j.gastro.2004.01.063. PMID 15168363
- [Background] Winther KV, Jess T, Langholz E, Munkholm P, Binder V. Survival and cause-specific mortality in ulcerative colitis: follow-up of a population-based cohort in Copenhagen County. Gastroenterology. 2003 Dec;125(6):1576-82. doi: 10.1053/j.gastro.2003.09.036. PMID 14724807
- [Background] Truelove SC, Pena AS. Course and prognosis of Crohn's disease. Gut. 1976 Mar;17(3):192-201. doi: 10.1136/gut.17.3.192. PMID 1269986
- [Background] Talbot RW, Heppell J, Dozois RR, Beart RW Jr. Vascular complications of inflammatory bowel disease. Mayo Clin Proc. 1986 Feb;61(2):140-5. doi: 10.1016/s0025-6196(12)65200-8. PMID 3080643
- [Background] Miehsler W, Reinisch W, Valic E, Osterode W, Tillinger W, Feichtenschlager T, Grisar J, Machold K, Scholz S, Vogelsang H, Novacek G. Is inflammatory bowel disease an independent and disease specific risk factor for thromboembolism? Gut. 2004 Apr;53(4):542-8. doi: 10.1136/gut.2003.025411. PMID 15016749
- [Background] Jackson LM, O'Gorman PJ, O'Connell J, Cronin CC, Cotter KP, Shanahan F. Thrombosis in inflammatory bowel disease: clinical setting, procoagulant profile and factor V Leiden. QJM. 1997 Mar;90(3):183-8. doi: 10.1093/qjmed/90.3.183. PMID 9093595
- [Background] Irving PM, Pasi KJ, Rampton DS. Thrombosis and inflammatory bowel disease. Clin Gastroenterol Hepatol. 2005 Jul;3(7):617-28. doi: 10.1016/s1542-3565(05)00154-0. PMID 16206491
- [Background] Solem CA, Loftus EV, Tremaine WJ, Sandborn WJ. Venous thromboembolism in inflammatory bowel disease. Am J Gastroenterol. 2004 Jan;99(1):97-101. doi: 10.1046/j.1572-0241.2003.04026.x. PMID 14687149